CLINICAL TRIAL: NCT05722795
Title: Use of Imatinib to Convert Triple Negative Breast Cancer Into ER-positive Breast Cancer
Brief Title: Use of Imatinib to Convert Triple Negative Breast Cancer Into ER-positive Breast Cancer (I-CONIC)
Acronym: I-CONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EudraCT 2020-005200-19
Record Dates: First submitted 2022-04-11; First posted 2023-02-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: Conversion of TNBC to Luminal BC
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Imatinib Mesylate; Tablets

STUDY DESIGN:
Intervention Model Description: Window-of-opportunity trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Short term Imatinib (Experimental): Imatinib 400 mg x 1 for 10 days before surgery.
  Interventions: Drug: Imatinib 400 MG Oral Tablet

INTERVENTIONS:
Drug: Imatinib 400 MG Oral Tablet — One tablet daily 10 days before surgery.
  Other Names: No other intervention

SUMMARY:
This is a single centre Window-of-Opportunity trial investigating the efficacy and feasibility of short term imatinib in patients with newly diagnosed triple negative breast cancer (TNBC) planned for surgery, with tumours ≥ 15 mm, any status in the axilla when neoadjuvant treatment not is considered as an option.

The primary aim is to determine the proportion of patients that converts to estrogen receptor (ER) positive breast cancer in the removed breast cancer tissue at surgery.

DETAILED DESCRIPTION:
This is a single centre Window-of-Opportunity trial that will investigate the efficacy and feasibility of short term (10 days) imatinib in patients with newly diagnosed TNBC planned for surgery, with tumours ≥ 15 mm, any status in the axilla and when neoadjuvant treatment not is considered as an option. Imatinib is given at a dose of 400 mg daily.

The primary aim is to determine the proportion of patients that converts to ER positive breast cancer in the removed breast cancer tissue at surgery.

The secondary aim is to evaluate the safety and adverse events (AE) will be collected throughout the study, from informed consent until 30 days after the last dose of the IMP imatinib.

AEs will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed invasive primary triple negative breast cancer≥15 mm) with any node status.
2. Age ≥18 years

   Triple Negative subtype is defined below:
   1. Hormone receptor status: the invasive tumour shall be ER- and progesterone receptor (PR) -negative [staining present in <10% by immunohistochemistry (IHC)].
   2. HER2 status: the invasive tumour shall be Human Epidermal growth factor Receptor (HER) 2-negative by the American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) guidelines
3. No previous systemic treatment for TNBC
4. No concurrent anti-cancer treatment. Treatment with Bisphosphonates may continue.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
6. Normal organ function as defined below:

   1. absolute white blood cell count ≥1.5 x 109/L
   2. platelets ≥100 x 109/L
   3. haemoglobin ≥90g/dL
   4. total bilirubin ≤1.5 x institutional upper normal limit (UNL)/dL (≤ 3 x UNL for patients with Gilbert´s syndrome)
   5. ASAT, ALAT, GGT and alkaline phosphatase levels < 1.5 × institutional UNL.
   6. albumin >2.5mg/dL
   7. Creatinine < 110 μmol/L
   8. T3, T4 and TSH (only patients with previous thyroid dysfunction)
7. Patients of childbearing potential must have a negative serum or urine pregnancy test within 8 days prior to start of imatinib treatment..

   Female patients of childbearing potential must agree to usecontraceptive methods with a failure rate below 1% per year during the study treatment and at least 90 days after the last dose of imatinib.
8. Patients must be able to take (swallow) an oral medication.
9. Patients must be capable to understand and comply with the protocol and has signed the informed consent.

Exclusion Criteria:

1. Patients suitable for neoadjuvant treatment.
2. Concomitant treatment for breast cancer within 14 days before registration.
3. Unable to adhere to the study procedures.
4. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, neurological conditions, physical examination or laboratory findings) that may interfere with the planned treatment or affect patient compliance.
5. Pregnancy and breast-feeding.
6. Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ).
7. Known human immunodeficiency virus (HIV) positivity.
8. Known active Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2029-06-28 (Estimated); Study Completion 2029-12-28 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of patients that convert to ER expressing breast cancer | From surgery of the first patient to up to 100 weeks thereafter.
  ER expression is determined by immunohistochemistry

SECONDARY OUTCOMES:
Adverse events | From time of the first included patient to up to 100 weeks thereafter.
  AEs are registered according to National Cancer Institute (NCI) CTCAE version 5.0.

OTHER OUTCOMES:
Exploratory analyses - gene expression profiles | From surgery of the first patient to up to 100 weeks thereafter.
  Gene expression profiles in tissue - biopsy and surgical specimen.
Exploratory analyses - gene expression profiles | From time of the first included patient to up to 100 weeks thereafter.
  Gene expression profiles determined in circulating tumour-DNA

CONTACTS AND LOCATIONS:
Overall Officials: Barbro K Linderholm, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Barbro Linderholm, Gothenburg, Sweden

REFERENCES:
- [Result] Roswall P, Bocci M, Bartoschek M, Li H, Kristiansen G, Jansson S, Lehn S, Sjolund J, Reid S, Larsson C, Eriksson P, Anderberg C, Cortez E, Saal LH, Orsmark-Pietras C, Cordero E, Haller BK, Hakkinen J, Burvenich IJG, Lim E, Orimo A, Hoglund M, Ryden L, Moch H, Scott AM, Eriksson U, Pietras K. Microenvironmental control of breast cancer subtype elicited through paracrine platelet-derived growth factor-CC signaling. Nat Med. 2018 May;24(4):463-473. doi: 10.1038/nm.4494. Epub 2018 Mar 12. PMID 29529015
- [Result] Jansson S, Aaltonen K, Bendahl PO, Falck AK, Karlsson M, Pietras K, Ryden L. The PDGF pathway in breast cancer is linked to tumour aggressiveness, triple-negative subtype and early recurrence. Breast Cancer Res Treat. 2018 Jun;169(2):231-241. doi: 10.1007/s10549-018-4664-7. Epub 2018 Jan 29. PMID 29380207
- [Result] Arnedos M, Roulleaux Dugage M, Perez-Garcia J, Cortes J. Window of Opportunity trials for biomarker discovery in breast cancer. Curr Opin Oncol. 2019 Nov;31(6):486-492. doi: 10.1097/CCO.0000000000000583. PMID 31464762